CLINICAL TRIAL: NCT03040154
Title: Engaging Immigrants in Preventive Parenting Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Joyce Javier, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCI-13-00159
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Health Behavior; Parenting; Social Acceptance
Keywords: Filipino
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Culturally-tailored video that includes parent testimonials, health and mental health clinicians, community-based providers, and church leaders
  Interventions: Other: Video Documentary entitled, "Para Sa Kinabukasan ng Mga Anak (For Our Children's Future)"
- Control Arm (Other): Usual care video publicly available describing the evidence-based parenting intervention
  Interventions: Other: Usual Care Video that is publicly available

INTERVENTIONS:
Other: Video Documentary entitled, "Para Sa Kinabukasan ng Mga Anak (For Our Children's Future)"
  Other Names: Intervention Arm
  Arms: Intervention Arm
Other: Usual Care Video that is publicly available
  Other Names: Control Arm
  Arms: Control Arm

SUMMARY:
The objective of this community-based randomized controlled trial is to evaluate the outcomes of a theory-based parent engagement intervention (i.e., culturally-tailored video) aimed at promoting the participation of Filipino parents and grandparents in an evidence-based preventive parenting intervention.

DETAILED DESCRIPTION:
Data will be obtained using pre and post surveys with self-report instruments and enrollment logs. It is hypothesized that 1) Parents and grandparents in the Intervention Arm will demonstrate greater behavioral outcomes (intention to enroll, actual enrollment, and participation in parenting intervention sessions) than those in the Control Arm. 2) Parents and grandparents in the Intervention Arm will show greater improvements from baseline in parent determinants (knowledge, beliefs, attitudes, benefits, and barriers) compared to the Control Arm. 3) Parents' intention to enroll, and actual enrollment in IY will be predicted by the study arm and parent determinants. This study is expected to have an important impact on the uptake of evidence-based parenting interventions among hard-to-reach populations and holds the promise of eliminating disparities in behavioral health outcomes in this understudied and growing minority population.

ELIGIBILITY:
Inclusion Criteria:

* The sample will consist of Filipino parents and grandparents of children/grandchildren between ages 6-12 years old. Inclusion criteria include:

  1. the parent or grandparent has at least one child between 6 to 12 years of age
  2. the participating parent/grandparent is Filipino
  3. At least one parent/grandparent is willing to complete pre and post surveys and watch a brief video
  4. the parent/grandparent is age 18 or older
  5. English fluency

Exclusion Criteria:

1. Younger than 18 years of age
2. Does not speak English
3. Target child has a developmental disability such as Trisomy 21 or autism
4. Parent or grandparent plans to move out of the area within the next nine months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R. Javier, MD, MPH, MS, Principal Investigator — Children's Hospital Los Angeles, University of Southern California Keck School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javier JR, Coffey DM, Palinkas LA, Kipke MD, Miranda J, Schrager SM. Promoting Enrollment in Parenting Programs Among a Filipino Population: A Randomized Trial. Pediatrics. 2019 Feb;143(2):e20180553. doi: 10.1542/peds.2018-0553. PMID 30679379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 595 participants were assessed for eligibility. Of these participants, 378 were excluded (221 did not meet inclusion criteria, 157 were not interested).
Pre-assignment Details: 217 participants were initially enrolled (i.e. they were CONSENTED and ASSIGNED to a group). Two participants dropped out before data was collected, which explains the changes from 217 participants who started to 215 participants who completed the study.
Groups:
- Intervention Arm: Culturally-tailored video that includes parent testimonials, health and mental health clinicians, community-based providers, and church leaders
  Video Documentary entitled, "Para Sa Kinabukasan ng Mga Anak (For Our Children's Future)"
- Control Arm: Usual care video publicly available describing the evidence-based parenting intervention
  Usual Care Video that is publicly available
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 110 | 105
Completed | 110 | 105
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 110 | 105 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing Values for Participant Age
  years
    number analyzed (Participants) | 109 | 103 | 212
    (all) | 45.93 (12.32) | 45.66 (11.12) | 45.80 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 86 | 164
  Male | 32 | 19 | 51
Relationship to Child [Count of Participants; unit: Participants]
  Biological Mother | 59 | 70 | 129
  Biological Father | 26 | 13 | 39
  Adpotive Father | 1 | 0 | 1
  Stepparent | 1 | 1 | 2
  Parent's Partner | 5 | 3 | 8
  Other Adult Relative | 2 | 4 | 6
  Other | 16 | 14 | 30
Marital Status [Count of Participants; unit: Participants]
  Never Married | 11 | 6 | 17
  Living Together | 2 | 1 | 3
  Married | 79 | 86 | 165
  Separated | 6 | 0 | 6
  Divorced | 7 | 8 | 15
  Widowed | 5 | 4 | 9
Child's Gender [Count of Participants; unit: Participants]
  Male | 51 | 50 | 101
  Female | 59 | 55 | 114
Income [Count of Participants; unit: Participants] — Population: Missing Values for Income
  Participants
    <20,00: number analyzed (Participants) | 110 | 103 | 213
    <20,00 | 29 | 20 | 49
    20,000-49,999: number analyzed (Participants) | 110 | 103 | 213
    20,000-49,999 | 42 | 31 | 73
    50,000-99,999: number analyzed (Participants) | 110 | 103 | 213
    50,000-99,999 | 28 | 36 | 64
    >100,00: number analyzed (Participants) | 110 | 103 | 213
    >100,00 | 11 | 16 | 27
Child's Birthplace [Count of Participants; unit: Participants]
  United States | 85 | 85 | 170
  Philippines | 22 | 20 | 42
  Other | 3 | 0 | 3
Education [Count of Participants; unit: Participants]
  Grades 0-8 | 1 | 0 | 1
  Grades 9-11 | 0 | 1 | 1
  High School or GED | 6 | 8 | 14
  Some College | 22 | 19 | 41
  College Graduate | 74 | 59 | 133
  Post-College Graduate | 7 | 18 | 25
Work Status [Count of Participants; unit: Participants]
  Full Time | 65 | 61 | 126
  Part Time | 21 | 13 | 34
  Working at Home | 2 | 5 | 7
  Looking for a Job | 6 | 14 | 20
  Not working by choice | 16 | 12 | 28
Parent's Birthplace [Count of Participants; unit: Participants]
  United States | 10 | 14 | 24
  Philippines | 99 | 90 | 189
  Other | 1 | 1 | 2
Primary Home Language [Count of Participants; unit: Participants]
  English | 44 | 47 | 91
  Tagalog | 40 | 35 | 75
  Ilocano | 2 | 5 | 7
  Bisaya | 6 | 1 | 7
  Other | 18 | 17 | 35
Child's Age [Mean (Standard Deviation); unit: years] — Population: Missing Values for Child's Age
  years
    number analyzed (Participants) | 109 | 104 | 213
    (all) | 8.73 (1.95) | 8.85 (2.05) | 8.79 (1.995)
Perceived Susceptibility to risky sexual activity [Mean (Full Range); unit: Units on a scale] — "Participating in Risky Sexual Activity"
  This measure asks parents to rate their child's chances of experiencing these problems on a scale of 0 to 100. Zero means you are certain your child will not experience this problem and 100 means that you are certain that he/she will experience the problem when he/she is a teenager. Population: Missing Values
  Total Median is "0" because most participants answered "0"
  Units on a scale
    number analyzed (Participants) | 109 | 101 | 210
    (all) | 6.68 [0 to 80] | 7.17 [0 to 70] | 6.91 [0 to 80]
Perceived Susceptibility to using illegal drugs [Mean (Full Range); unit: units on a scale] — "Occasionally using illegal drugs"
  This measure asks parents to rate their child's chances of experiencing these problems on a scale of 0 to 100. Zero means you are certain your child will not experience this problem and 100 means that you are certain that he/she will experience the problem when he/she is a teenager. Population: Data missing for some participants
  units on a scale
    number analyzed (Participants) | 110 | 101 | 211
    (all) | 4.2455 [0 to 80.00] | 5.4257 [0 to 91.00] | 4.8104 [0 to 91.00]
Perceived Susceptibility to thoughts of suicide [Mean (Full Range); unit: units on a scale] — "Having thoughts about suicide"
  This measure asks parents to rate their child's chances of experiencing these problems on a scale of 0 to 100. Zero means you are certain your child will not experience this problem and 100 means that you are certain that he/she will experience the problem when he/she is a teenager. Population: Data missing for some participants
  units on a scale
    number analyzed (Participants) | 110 | 101 | 211
    (all) | 4.4091 [0 to 51.00] | 4.8812 [0 to 60.00] | 4.6351 [0 to 60]
Knowledge of Filipino mental health disparities: Suicide [Mean (Full Range); unit: units on a scale] — "Filipino teenagers in the US are at higher risk of having suicidal thoughts compared to other ethnic groups in the US"
  This measure asks about knowledge of Filipino mental health disparities, specifically suicide, using a 7-point likert scale where 1= strongly disagree, 2=disagree, 3=disagree a little, 4= neutral, 5=agree a little, 6=agree, 7=strongly agree. Population: Data missing for some participants
  units on a scale
    number analyzed (Participants) | 110 | 104 | 214
    (all) | 2.39 [1.0 to 4.0] | 2.45 [1.0 to 5.0] | 2.42 [1.0 to 5.0]
Knowledge of Filipino behavioral health disparities: drug use [Mean (Full Range); unit: units on a scale] — "Filipino teenagers in the US have higher rates of alcohol and drug use compared with other Asian subgroups"
  This measure asks about knowledge of Filipino behavioral health disparities, specifically alcohol and drug use, using a 7-point likert scale where 1= strongly disagree, 2=disagree, 3=disagree a little, 4= neutral, 5=agree a little, 6=agree, 7=strongly agree Population: Data missing for some participants
  units on a scale
    number analyzed (Participants) | 110 | 104 | 214
    (all) | 2.75 [1.0 to 5.0] | 2.86 [1.0 to 5.0] | 2.8 [1.0 to 5.0]

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in Evidence-Based Parenting Program
Description: The number of participants from each arm who enrolled in the Incredible Years Parenting Program after completing this study. Enrollment in the parenting program helped determine if the culturally-tailored video intervention effectively increases program participation among Filipino parents.
Time Frame: Up to two years after completing the survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 110 | 105
Participants | 27 | 12
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.33 to 5.35]

ADVERSE EVENTS:
Time Frame: Through study completion, for up to 6 months
Arm/Group | Intervention Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/105
Other Adverse Events (participants affected / at risk) | 0/110 | 0/105

LIMITATIONS AND CAVEATS:
This was conducted in urban populations of Filipinos in Southern California, so findings may not generalize to non-urban or other racial/ethnic populations. Knowledge and susceptibility were also self-reported and subject to social desirability bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No